CLINICAL TRIAL: NCT05775926
Title: The Effect of Training Given to Nurses Caring for Dying Cancer Patients and Their Families on Care and Difficulties
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Meltem Akbaş, Assistant Professor, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 05.04.2019/87
Record Dates: First submitted 2023-02-22; First posted 2023-03-20 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Dying Patient; Nursing Caries
Keywords: Nursing care; Dying patient; Cancer
MeSH Terms: conditions — Neoplasms | interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Experimental Group: Nurses who met the criteria for participating in the study were informed about the study and their consent was obtained. Data collection forms were collected by the researcher at the end of the working hours. Training groups were formed on the days and times determined according to the interviews with the clinics where the research was conducted. In each hospital, training groups were formed outside the working hours of the nurses. The training was given to the nurses in the intervention group in an environment suitable for training in two days and 4 modules using interactive teaching methods. After the training, a month was waited for the nurses in the intervention group to experience care. One month after the training was given, data collection forms were distributed to the nurses in the intervention group and asked to fill in according to their self-reports.
  Interventions: Other: Education
- Control (No Intervention): Control Group: Nurses who met the criteria for participating in the study were informed about the study and their consent was obtained. Data collection forms were collected by the researcher at the end of the working hours. No training was given to the control group. However, after the post-test application was made to the control group, the same training was given to the experimental group. One month later, data collection forms were distributed to the nurses in the control group and they were asked to fill in according to their self-reports. Data collection forms were collected by the researcher at the end of the working hours. Filling in the data takes about 15 minutes.

INTERVENTIONS:
Other: Education — Nursing Care and Challenges Training for Nurses Caring for Dying Cancer Patients and Their Families was given in 4 modules and 2 days.
  Arms: Experimental

SUMMARY:
Nursing is a profession that is human and is based on nursing care. Humans are social creatures that need care from the moment they are born.Today's scientific developments and changing technology have affected the health system.Many dying patients want to be hospitalized in order to receive better care and treatment. Depending on this situation, the frequency of nurses giving care to dying patients and their families has increased in hospitals. In order to increase the quality of the care given to the dying patient and his family and to reduce the difficulties experienced while giving this care, the nurse who provides the care should have sufficient knowledge and skills about the care of the dying patient and his family.

This research will be conducted as a randomized controlled experimental study in order to determine the effect of education on the nursing care given and the difficulties experienced by the nurses who care for the dying cancer patients and their families.

DETAILED DESCRIPTION:
The research was carried out to determine the effect of the training given to the nurses who care for the dying cancer patients and their families, on the nursing care and the difficulties experienced.

H1: There is a significant difference between the "Nursing Care Scale for Dying Patients and Their Families" pre- and post-test scores of the intervention and control groups.

H2: There is a significant difference between the pre-test and post-test scores of the "Nurse Difficulty Scale for Dying Patients and Their Families" of the intervention and control groups.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer
* Working in a clinic where adult cancer patients are hospitalized for at least 1 year

Exclusion Criteria:

* On leave
* Not volunteering

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
The Nursing Care Scale for Dying Patients and Their Families [NCD] | 1 month
  While the score to be obtained from each of the sub-dimensions of the scale varies between 3-15, the total score is between 15-60. The higher the score obtained from the scale, the higher the quality of nursing care.
The Nurse's Difficulty Scale for Dying Patients and Their Families [NDD] | 1 month
  While the score to be obtained from each of the sub-dimensions of the scale varies between 3-15, the total score is between 15-60. As the score obtained from the scale increases, the difficulties experienced by the nurses increase.

CONTACTS AND LOCATIONS:
Overall Officials: Meltem Akbaş, PhD, Principal Investigator — Cukurova University
Locations (1):
- Cukurova University, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No